CLINICAL TRIAL: NCT03861767
Title: Randomized, Embedded, Multifactorial, Adaptive Platform Trial for Optimizing Surgical Outcomes at UPMC
Brief Title: REMAP Trial for Optimizing Surgical Outcomes at UPMC
Acronym: UPMCREMAP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not enough enrollment due to the COVID19 pandemic.
Sponsor: Matthew Neal MD (Other)
Collaborators: University of Pittsburgh Medical Center (Other); Berry Consultants (Other)
Responsible Party: Sponsor-Investigator, Matthew Neal MD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY19090186
Record Dates: First submitted 2019-01-21; First posted 2019-03-04 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Aging
Keywords: Prehabilitation
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- SPRY: Metformin LD-SC (low-dose, short course) (Experimental): LD-SC (low-dose, short course)
  Participants take Metformin ER 500 mg daily for 7-28 days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Interventions: Drug: Metformin ER
- SPRY: Metformin LD-IC (low-dose, intermediate course) (Experimental): LD-IC (low-dose, intermediate course)
  Participants take Metformin ER 500 mg daily for 29-90 days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Interventions: Drug: Metformin ER
- SPRY: Metformin LD-LC (low-dose, long course) (Experimental): LD-LC (low-dose, long course)
  Participants take Metformin ER 500 mg daily for 90+ days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Interventions: Drug: Metformin ER
- SPRY: Metformin ID-SC (intermediate-dose, short course) (Experimental): ID-SC (intermediate-dose, short course)
  Participants take Metformin ER 1000 mg daily for 7-28 days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Interventions: Drug: Metformin ER
- SPRY: Metformin ID-IC (intermediate-dose, intermediate course) (Experimental): ID-IC (intermediate-dose, intermediate course)
  Participants take Metformin ER 1000 mg daily for 29-90 days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Interventions: Drug: Metformin ER
- SPRY: Metformin ID-LC (intermediate-dose, long course) (Experimental): ID-LC (intermediate-dose, long course)
  Participants take Metformin ER 1000 mg daily for 90+ days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Interventions: Drug: Metformin ER
- SPRY: Metformin HD-SC (high-dose, short course) (Experimental): HD-SC (high-dose, short course)
  After a 7 day run-in of Metformin ER 1000 mg, participants take Metformin ER 1500 mg daily for 7-28 days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Interventions: Drug: Metformin ER
- SPRY: Metformin HD-IC (high-dose, intermediate course) (Experimental): HD-IC (high-dose, intermediate course)
  After a 7 day run-in of Metformin ER 1000 mg, participants take Metformin ER 1500 mg daily for 29-90 days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Interventions: Drug: Metformin ER
- SPRY: Metformin HD-LC (high-dose, long course) (Experimental): HD-LC (high-dose, long course)
  After a 7 day run-in of Metformin ER 1000 mg, participants take Metformin ER 1500 mg daily for 90+ days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Interventions: Drug: Metformin ER
- SPRY: Placebo (Placebo Comparator): Participants are randomized to receive dose matched placebo to take daily for either short-, intermediate-, or long-course.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin ER — tablet
  Other Names: Metformin Extended Release
  Arms: SPRY: Metformin HD-IC (high-dose, intermediate course); SPRY: Metformin HD-LC (high-dose, long course); SPRY: Metformin HD-SC (high-dose, short course); SPRY: Metformin ID-IC (intermediate-dose, intermediate course); SPRY: Metformin ID-LC (intermediate-dose, long course); SPRY: Metformin ID-SC (intermediate-dose, short course); SPRY: Metformin LD-IC (low-dose, intermediate course); SPRY: Metformin LD-LC (low-dose, long course); SPRY: Metformin LD-SC (low-dose, short course)
Drug: Placebo — Matched placebo in doses of 1, 2 and 3 tablets to coincide with the 500, 1000, and 1500 mg arms.
  Arms: SPRY: Placebo

SUMMARY:
The purpose of this project is to determine the effect of various interventions to improve patient outcome as defined by hospital free days at day 90 for adult patients undergoing elective surgery. Within this project, multiple studies may be conducted.

The structure of this project permits:

* the testing of multiple treatments at the same time within the same patient
* the use of early study results to provide better treatment options to future patients
* the removal of treatments which are shown to be less effective than the other treatments
* the addition of new treatments

The first study to be conducted under this project (IRB STUDY19090186) is the Strategies to Promote ResiliencY (SPRY) clinical trial (IRB PRO18060038).

The SPRY clinical trial will determine the effectiveness of Metformin on improving surgical outcomes among nondiabetic older adults who are scheduled for elective surgery.

ELIGIBILITY:
UPMC REMAP

Inclusion Criteria:

* Adult patient evaluated pre-operatively for elective surgery at UPMC
* Minimum lead time before surgery to provide domain specific intervention (range 7-180 days pre-operatively)
* Age greater to or equal to 18 years of age

Exclusion Criteria:

* Death is deemed to be imminent or inevitable
* Emergency surgical procedure without suitable lead-in time
* Previous participation in this REMAP within the last 90 days, flagged by elective or emergency surgical encounter at UPMC in the past 90 days

SPRY Domain

Inclusion Criteria:

* Age >= 60 years
* Age < 60 but evidence of comorbidity risk as represented by a Charlson Comorbidity Index of > 2 in 12 months prior to enrollment
* Able to take an oral medication in non-crushable pill form
* Women must be post-menopausal, which is defined as not having a menstrual period within the last 12 months

Exclusion Criteria:

* The treating clinician believes that participation in the domain would not be in the best interest of the patient
* Pre-existing diabetes type I or II
* Women of child-bearing potential
* Hospital stay <24 hours
* Presently taking metformin or prior use in the past 6 months
* Evidence of an absolute or relative contraindication to Metformin therapy

  * Known allergy to metformin
  * Acute or chronic metabolic acidosis with or without coma
  * Hemodialysis, end-stage renal disease, or Glomerular Filtration Rate (GFR) < 45 in the prior 30 days
  * Ongoing treatment with therapy known to have significant drug-drug interaction with metformin (carbonic anhydrase inhibitors, cimetidine, gliptins)
  * History of lactic acidosis
  * History of excessive alcohol intake
  * Severe hepatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Neal, MD, FACS, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data underlying the results reported in journal articles, subject to appropriate security controls, may be available for sharing with other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Relevant data may be available 1 year following publication
Access Criteria: Data access is subject to a methodologically sound proposal and the necessary data sharing agreements.

REFERENCES:
- [Derived] Reitz KM, Seymour CW, Vates J, Quintana M, Viele K, Detry M, Morowitz M, Morris A, Methe B, Kennedy J, Zuckerbraun B, Girard TD, Marroquin OC, Esper S, Holder-Murray J, Newman AB, Berry S, Angus DC, Neal M. Strategies to Promote ResiliencY (SPRY): a randomised embedded multifactorial adaptative platform (REMAP) clinical trial protocol to study interventions to improve recovery after surgery in high-risk patients. BMJ Open. 2020 Sep 29;10(9):e037690. doi: 10.1136/bmjopen-2020-037690. PMID 32994242

RESULTS

PARTICIPANT FLOW:
Groups:
- SPRY: Metformin LD-SC (Low-dose, Short Course): LD-SC (low-dose, short course)
  Participants take Metformin ER 500 mg daily for 7-28 days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Metformin ER: tablet
- SPRY: Metformin LD-IC (Low-dose, Intermediate Course): LD-IC (low-dose, intermediate course)
  Participants take Metformin ER 500 mg daily for 29-90 days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Metformin ER: tablet
- SPRY: Metformin LD-LC (Low-dose, Long Course): LD-LC (low-dose, long course)
  Participants take Metformin ER 500 mg daily for 90+ days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Metformin ER: tablet
- SPRY: Metformin ID-SC (Intermediate-dose, Short Course): ID-SC (intermediate-dose, short course)
  Participants take Metformin ER 1000 mg daily for 7-28 days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Metformin ER: tablet
- SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course): ID-IC (intermediate-dose, intermediate course)
  Participants take Metformin ER 1000 mg daily for 29-90 days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Metformin ER: tablet
- SPRY: Metformin ID-LC (Intermediate-dose, Long Course): ID-LC (intermediate-dose, long course)
  Participants take Metformin ER 1000 mg daily for 90+ days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Metformin ER: tablet
- SPRY: Metformin HD-SC (High-dose, Short Course): HD-SC (high-dose, short course)
  After a 7 day run-in of Metformin ER 1000 mg, participants take Metformin ER 1500 mg daily for 7-28 days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Metformin ER: tablet
- SPRY: Metformin HD-IC (High-dose, Intermediate Course): HD-IC (high-dose, intermediate course)
  After a 7 day run-in of Metformin ER 1000 mg, participants take Metformin ER 1500 mg daily for 29-90 days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Metformin ER: tablet
- SPRY: Metformin HD-LC (High-dose, Long Course): HD-LC (high-dose, long course)
  After a 7 day run-in of Metformin ER 1000 mg, participants take Metformin ER 1500 mg daily for 90+ days prior to their elective surgical procedure as determined by the patient's scheduling of their surgery. Participants take this same dose of Metformin ER for 90 days after their surgical procedure.
  Metformin ER: tablet
Period: Overall Study
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Started | 39 | 20 | 5 | 39 | 19 | 8 | 40 | 26 | 0 | 106
Underwent Surgery | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Drug Compliance | 34 | 19 | 4 | 37 | 15 | 8 | 35 | 21 | 0 | 95
Completed (This total number is for intention-to-treat group. Per-Protocol group is the compliant group - (the group that did not undergo surgery + group that withdrew)) | 37 | 19 | 5 | 34 | 17 | 7 | 37 | 25 | 0 | 101
Not Completed | 2 | 1 | 0 | 5 | 2 | 1 | 3 | 1 | 0 | 5
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 5 | 2 | 1 | 3 | 1 | 0 | 5

BASELINE CHARACTERISTICS:
Population: None of the participants were randomized to the high-dose long course combination of drug dose and preoperative duration.
Groups:
- Total: Total of all reporting groups
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo | Total
Number analyzed (Participants) | 39 | 20 | 5 | 39 | 19 | 8 | 40 | 26 | 0 | 106 | 302
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 4 | 0 | 16 | 7 | 1 | 14 | 3 | 0 | 37 | 95
  >=65 years | 26 | 16 | 5 | 23 | 12 | 7 | 26 | 23 | 0 | 69 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (6.9) | 69.0 (6.1) | 70.8 (5.1) | 67.7 (7.3) | 68.6 (8.4) | 71.1 (5.8) | 67.5 (8.2) | 70.2 (6.5) |  | 67.8 (5.7) | 68.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 8 | 3 | 17 | 8 | 2 | 11 | 14 | 0 | 50 | 134
  Male | 18 | 12 | 2 | 22 | 11 | 6 | 29 | 12 | 0 | 56 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 38 | 19 | 4 | 37 | 19 | 8 | 39 | 25 | 0 | 106 | 295
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 4 | 1 | 0 | 1 | 3 | 0 | 5 | 15
  White | 38 | 17 | 4 | 33 | 18 | 8 | 39 | 21 | 0 | 101 | 279
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.9 (5.5) | 30.9 (4.7) | 31.3 (4.2) | 30.9 (5.9) | 28.0 (4.6) | 26.2 (5.1) | 30.5 (10.7) | 30.6 (6.6) |  | 30.2 (6.4) | 30.3 (6.7)
Risk analysis index score [Mean (Standard Deviation); unit: units on a scale] — This is a measure of frailty. Score is prospectively calculated during the preoperative visit and is a score that ranges from 0-81. A higher score represents increased frailty and higher susceptibility to postoperative complications.
  units on a scale | 27.2 (6.9) | 25.2 (5.9) | 31.0 (13.5) | 25.6 (5.5) | 22.8 (3.5) | 24.2 (2.3) | 25.5 (7.4) | 26.1 (4.6) |  | 25.8 (6.4) | 25.8 (6.3)
Smoking status [Count of Participants; unit: Participants]
  Active | 1 | 3 | 0 | 6 | 0 | 1 | 2 | 1 | 0 | 7 | 21
  Quit | 15 | 4 | 2 | 17 | 6 | 2 | 18 | 10 | 0 | 48 | 122
  Never | 23 | 13 | 2 | 16 | 13 | 5 | 19 | 15 | 0 | 50 | 156
  Unknown status | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
History of Stroke [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 4 | 11
  No | 38 | 20 | 3 | 37 | 17 | 8 | 40 | 26 | 0 | 102 | 291
History of chronic obstructive pulmonary disease [Count of Participants; unit: Participants]
  Yes | 1 | 1 | 1 | 5 | 0 | 1 | 3 | 5 | 0 | 12 | 29
  No | 38 | 19 | 4 | 34 | 19 | 7 | 37 | 21 | 0 | 94 | 273
History of coronary artery disease [Count of Participants; unit: Participants]
  Yes | 6 | 2 | 0 | 4 | 3 | 1 | 6 | 4 | 0 | 15 | 41
  No | 33 | 18 | 5 | 35 | 16 | 7 | 34 | 22 | 0 | 91 | 261
History of congestive heart failure [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 5
  No | 38 | 20 | 5 | 38 | 19 | 8 | 39 | 26 | 0 | 104 | 297
Surgical strata [Count of Participants; unit: Participants]
  No operation | 3 | 0 | 0 | 4 | 0 | 0 | 2 | 3 | 0 | 8 | 20
  Spine surgery | 10 | 6 | 1 | 9 | 3 | 1 | 12 | 6 | 0 | 34 | 82
  General surgery/Oncological surgery | 13 | 9 | 3 | 10 | 10 | 5 | 12 | 12 | 0 | 33 | 107
  Colorectal surgery | 2 | 3 | 1 | 4 | 5 | 0 | 6 | 2 | 0 | 13 | 36
  Other | 11 | 2 | 0 | 12 | 1 | 2 | 8 | 3 | 0 | 18 | 57

OUTCOME MEASURES:

1. Primary Outcome: Hospital Free Days (HFD)
Description: 90 - the number of days during the index stay minus the number of days readmitted during the 90 days after surgery. Death within 90 days after surgery is recorded as -1 HFD.
Time Frame: Day 90 from the date of the elective surgical procedure
Population: Participants were analyzed using intention-to-treat analysis. Participants that did not undergo an operation were excluded.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Days | 87 [84.8 to 89.2] | 88.5 [86.8 to 90] | 85 [84 to 85] | 88 [85 to 90] | 88 [86.5 to 90] | 89.5 [89 to 90] | 88 [85 to 90] | 87 [84 to 90] |  | 87 [85 to 90]
Statistical Analysis 1: Comparison: SPRY: Metformin LD-SC (Low-dose, Short Course) vs SPRY: Metformin LD-IC (Low-dose, Intermediate Course) vs SPRY: Metformin LD-LC (Low-dose, Long Course) vs SPRY: Placebo; Low dose groups collapsed and compared to placebo; Test type: Superiority; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.67 to 1.97]
Statistical Analysis 2: Comparison: SPRY: Metformin ID-SC (Intermediate-dose, Short Course) vs SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) vs SPRY: Metformin ID-LC (Intermediate-dose, Long Course) vs SPRY: Placebo; Intermediate dose groups were collapsed and compared to placebo; Test type: Superiority; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.42 to 1.25]
Statistical Analysis 3: Comparison: SPRY: Metformin HD-SC (High-dose, Short Course) vs SPRY: Metformin HD-IC (High-dose, Intermediate Course) vs SPRY: Placebo; High dose groups were collapsed and compared to placebo; Test type: Superiority; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.61 to 1.84]

2. Secondary Outcome: Incidence of ICU Admission After Surgery
Description: The intended measure of this outcome is to get the rate of ICU admission per described group or the number of participants that had an ICU admission within each group.
Time Frame: Participants will be followed for the duration of their hospital admission, estimated to be 2-4 days in the event ICU admission is needed
Population: Participants analyzed using intention-to-treat analysis. Participants that did not undergo surgery were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Participants | 3 | 2 | 0 | 3 | 2 | 1 | 3 | 1 | 0 | 10
Statistical Analysis 1: Comparison: SPRY: Metformin LD-SC (Low-dose, Short Course) vs SPRY: Metformin LD-IC (Low-dose, Intermediate Course) vs SPRY: Metformin LD-LC (Low-dose, Long Course) vs SPRY: Metformin ID-SC (Intermediate-dose, Short Course) vs SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) vs SPRY: Metformin ID-LC (Intermediate-dose, Long Course) vs SPRY: Metformin HD-SC (High-dose, Short Course) vs SPRY: Metformin HD-IC (High-dose, Intermediate Course) vs SPRY: Placebo; All intervention groups were grouped together and compared to placebo; Test type: Superiority; p = 0.92, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.52 to 2.03]

3. Secondary Outcome: Incidence and Total Number of Reoperation/Reintervention
Description: This outcome is also intended to measure the rate of Reoperation/reintervention within each group or the total number of participants that had a Reoperation/reintervention within each group as shown below
Time Frame: Day 90 from the date of the elective surgical procedure
Population: Participants were analyzed using intention-to-trial analysis. Participants that did not undergo an operation were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Participants | 8 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 14
Statistical Analysis 1: Comparison: SPRY: Metformin LD-SC (Low-dose, Short Course) vs SPRY: Metformin LD-IC (Low-dose, Intermediate Course) vs SPRY: Metformin LD-LC (Low-dose, Long Course) vs SPRY: Metformin ID-SC (Intermediate-dose, Short Course) vs SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) vs SPRY: Metformin ID-LC (Intermediate-dose, Long Course) vs SPRY: Metformin HD-SC (High-dose, Short Course) vs SPRY: Metformin HD-IC (High-dose, Intermediate Course) vs SPRY: Placebo; All intervention groups were grouped together and compared to placebo; Test type: Superiority; p = 0.80, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.52 to 2.00]

4. Secondary Outcome: Venous Thromboembolic Events Including Deep Vein Thrombosis and Pulmonary Embolism
Description: The intended measure from this outcome is to also show the rate of Venous thromboembolic events or the number of participants with Venous thromboembolic events within each group
Time Frame: Day 90 from the date of the elective surgical procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Participants | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Statistical Analysis 1: Comparison: SPRY: Metformin LD-SC (Low-dose, Short Course) vs SPRY: Metformin LD-IC (Low-dose, Intermediate Course) vs SPRY: Metformin LD-LC (Low-dose, Long Course) vs SPRY: Metformin ID-SC (Intermediate-dose, Short Course) vs SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) vs SPRY: Metformin ID-LC (Intermediate-dose, Long Course) vs SPRY: Metformin HD-SC (High-dose, Short Course) vs SPRY: Metformin HD-IC (High-dose, Intermediate Course) vs SPRY: Placebo; All intervention groups were grouped together and compared to placebo; Test type: Superiority; p = 0.65, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.49 to 3.11]

5. Secondary Outcome: Number of Participants With Surgical Site Infection
Time Frame: Day 30 from the date of the elective surgical procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Participants | 2 | 2 | 1 | 3 | 0 | 0 | 1 | 2 | 0 | 4
Statistical Analysis 1: Comparison: SPRY: Metformin LD-SC (Low-dose, Short Course) vs SPRY: Metformin LD-IC (Low-dose, Intermediate Course) vs SPRY: Metformin LD-LC (Low-dose, Long Course) vs SPRY: Metformin ID-SC (Intermediate-dose, Short Course) vs SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) vs SPRY: Metformin ID-LC (Intermediate-dose, Long Course) vs SPRY: Metformin HD-SC (High-dose, Short Course) vs SPRY: Metformin HD-IC (High-dose, Intermediate Course) vs SPRY: Placebo; All intervention groups were grouped together and compared to placebo; Test type: Superiority; p = 0.23, Regression, Logistic; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.73 to 3.62]

6. Secondary Outcome: Number of Participants With Surgical Site Occurrence
Time Frame: Day 30 from the date of the elective surgical procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Participants | 3 | 2 | 1 | 3 | 0 | 0 | 5 | 5 | 0 | 8
Statistical Analysis 1: Comparison: SPRY: Metformin LD-SC (Low-dose, Short Course) vs SPRY: Metformin LD-IC (Low-dose, Intermediate Course) vs SPRY: Metformin LD-LC (Low-dose, Long Course) vs SPRY: Metformin ID-SC (Intermediate-dose, Short Course) vs SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) vs SPRY: Metformin ID-LC (Intermediate-dose, Long Course) vs SPRY: Metformin HD-SC (High-dose, Short Course) vs SPRY: Metformin HD-IC (High-dose, Intermediate Course) vs SPRY: Placebo; All intervention groups were grouped together and compared to placebo; Test type: Superiority; p = 0.31, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.71 to 2.86]

7. Secondary Outcome: Organ Failure Free Days
Time Frame: Day 30 from the date of the elective surgical procedure
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Days
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Days | 29.84 (0.53) | 29.93 (0.22) | 29.97 (0.03) | 29.96 (0.04) | 29.86 (0.32) | 29.98 (0.02) | 29.88 (0.50) | 29.94 (0.21) |  | 29.90 (0.27)
Statistical Analysis 1: Comparison: SPRY: Metformin LD-SC (Low-dose, Short Course) vs SPRY: Metformin LD-IC (Low-dose, Intermediate Course) vs SPRY: Metformin LD-LC (Low-dose, Long Course) vs SPRY: Metformin ID-SC (Intermediate-dose, Short Course) vs SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) vs SPRY: Metformin ID-LC (Intermediate-dose, Long Course) vs SPRY: Metformin HD-SC (High-dose, Short Course) vs SPRY: Metformin HD-IC (High-dose, Intermediate Course) vs SPRY: Placebo; All intervention groups were grouped together and compared to placebo; Test type: Superiority; p = 0.97, Regression, Linear; Beta-coefficient = 0.0011, Standard Error of Mean 0.042

8. Secondary Outcome: Hospital Length of Stay (LOS)
Time Frame: Participants will be followed for the duration of their hospital admission, estimated to be 2-4 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Days | 3.9 (4.9) | 2.5 (2.8) | 4.00 (2.3) | 3.6 (4.1) | 2.6 (3.4) | 0.4 (0.5) | 4.3 (6.7) | 3.3 (3.2) |  | 4.2 (7.4)
Statistical Analysis 1: Comparison: SPRY: Metformin LD-SC (Low-dose, Short Course) vs SPRY: Metformin LD-IC (Low-dose, Intermediate Course) vs SPRY: Metformin LD-LC (Low-dose, Long Course) vs SPRY: Metformin ID-SC (Intermediate-dose, Short Course) vs SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) vs SPRY: Metformin ID-LC (Intermediate-dose, Long Course) vs SPRY: Metformin HD-SC (High-dose, Short Course) vs SPRY: Metformin HD-IC (High-dose, Intermediate Course) vs SPRY: Placebo; All intervention groups were grouped together and compared to placebo; Test type: Superiority; p = 0.30, Regression, Linear; Beta-coefficient = -0.76, Standard Error of Mean 0.74

9. Secondary Outcome: ICU (Intensive Care Unit) Length of Stay (LOS)
Time Frame: Participants will be followed for the duration of their hospital admission, estimated to be 2-4 days, in the event admission to an ICU is needed
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Days | 0.1 (0.4) | 0.3 (0.9) | 0.0 (0.0) | 0.3 (1.3) | 0.3 (0.9) | 0.1 (0.3) | 0.1 (0.6) | 0.1 (0.5) |  | 0.2 (0.7)
Statistical Analysis 1: Comparison: SPRY: Metformin LD-SC (Low-dose, Short Course) vs SPRY: Metformin LD-IC (Low-dose, Intermediate Course) vs SPRY: Metformin LD-LC (Low-dose, Long Course) vs SPRY: Metformin ID-SC (Intermediate-dose, Short Course) vs SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) vs SPRY: Metformin ID-LC (Intermediate-dose, Long Course) vs SPRY: Metformin HD-SC (High-dose, Short Course) vs SPRY: Metformin HD-IC (High-dose, Intermediate Course) vs SPRY: Placebo; All intervention groups were grouped together and compared to placebo; Test type: Superiority; p = 0.65, Regression, Linear; Beta-coefficient = 0.27, Standard Error of Mean 0.59

10. Secondary Outcome: Mortality
Time Frame: Day 90 from the date of the elective surgical procedure
Population: Participants were analyzed using intention-to-trial analysis. Participants that did not undergo an operation were excluded. Only one mortality was observed and thus no statistical analysis was performed
Measure: Count of Participants; unit: Participants
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Participants | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Hospital Readmission Rate
Time Frame: Day 90 from the date of the elective surgical procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Participants | 5 | 2 | 1 | 6 | 3 | 0 | 5 | 0 | 0 | 9
Statistical Analysis 1: Comparison: SPRY: Metformin LD-SC (Low-dose, Short Course) vs SPRY: Metformin LD-IC (Low-dose, Intermediate Course) vs SPRY: Metformin LD-LC (Low-dose, Long Course) vs SPRY: Metformin ID-SC (Intermediate-dose, Short Course) vs SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) vs SPRY: Metformin ID-LC (Intermediate-dose, Long Course) vs SPRY: Metformin HD-SC (High-dose, Short Course) vs SPRY: Metformin HD-IC (High-dose, Intermediate Course) vs SPRY: Placebo; Test type: Superiority; p = 0.27, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.74 to 2.86]

12. Secondary Outcome: Gastrointestinal Intolerance
Time Frame: From enrollment to day 90 after surgery
Population: All participants included. Group with zero participants added for completion
Measure: Count of Participants; unit: Participants
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 39 | 20 | 5 | 39 | 19 | 8 | 40 | 26 | 0 | 106
Participants | 7 | 4 | 1 | 4 | 5 | 0 | 6 | 3 | 0 | 6
Statistical Analysis 1: Comparison: SPRY: Metformin LD-SC (Low-dose, Short Course) vs SPRY: Metformin LD-IC (Low-dose, Intermediate Course) vs SPRY: Metformin LD-LC (Low-dose, Long Course) vs SPRY: Metformin ID-SC (Intermediate-dose, Short Course) vs SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) vs SPRY: Metformin ID-LC (Intermediate-dose, Long Course) vs SPRY: Metformin HD-SC (High-dose, Short Course) vs SPRY: Metformin HD-IC (High-dose, Intermediate Course) vs SPRY: Placebo; All intervention groups were collapsed and compared to placebo; Test type: Superiority; p = 0.01, Regression, Logistic; Odds Ratio (OR) = 2.98, 95% CI 2-sided [1.19 to 7.44]

13. Secondary Outcome: SAE (Serious Adverse Event) as Defined in Core Protocol (Mild, Moderate, Severe, Life Threatening/Disabling; Adjudicated as Related, Possibly Related, Unrelated)
Description: The number of participants here includes the full cohort because adverse events were recorded for all participants while other outcome measures were only recorded for participants that underwent surgery
Time Frame: From enrollment to day 90 after surgery
Population: All participants included. Group with zero participants included for completion
Measure: Count of Participants; unit: Participants
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 39 | 20 | 5 | 39 | 19 | 8 | 40 | 26 | 0 | 106
Participants
  Mild - related | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 2
  Mild- possibly related | 3 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 4
  Mild - unrelated | 5 | 2 | 2 | 5 | 1 | 1 | 2 | 0 | 0 | 3
  Moderate - related | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Moderate- possibly related | 4 | 1 | 0 | 1 | 0 | 0 | 5 | 2 | 0 | 0
  Moderate - unrelated | 1 | 2 | 0 | 1 | 2 | 0 | 4 | 1 | 0 | 3
  Severe - related | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe- possibly related | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe - unrelated | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
  life threatening/disabling - related | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  life threatening/disabling - possibly related | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  life threatening/disabling - unrelated | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: SPRY: Metformin LD-SC (Low-dose, Short Course) vs SPRY: Metformin LD-IC (Low-dose, Intermediate Course) vs SPRY: Metformin LD-LC (Low-dose, Long Course) vs SPRY: Metformin ID-SC (Intermediate-dose, Short Course) vs SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) vs SPRY: Metformin ID-LC (Intermediate-dose, Long Course) vs SPRY: Metformin HD-SC (High-dose, Short Course) vs SPRY: Metformin HD-IC (High-dose, Intermediate Course) vs SPRY: Placebo; All intervention groups were collapsed and compared to placebo; Test type: Superiority; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 2.67, 95% CI 2-sided [1.34 to 5.30]

14. Secondary Outcome: Discharge Disposition
Time Frame: as for outcome 9
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Participants
  Home | 29 | 18 | 5 | 30 | 17 | 7 | 33 | 18 | 0 | 85
  Skilled nursing facility/Rehabilitation facility | 5 | 1 | 0 | 1 | 0 | 0 | 2 | 4 | 0 | 8
  Death/Hospice | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing data | 2 | 1 | 0 | 4 | 2 | 1 | 3 | 1 | 0 | 5
Statistical Analysis 1: Comparison: SPRY: Metformin LD-SC (Low-dose, Short Course) vs SPRY: Metformin LD-IC (Low-dose, Intermediate Course) vs SPRY: Metformin LD-LC (Low-dose, Long Course) vs SPRY: Metformin ID-SC (Intermediate-dose, Short Course) vs SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) vs SPRY: Metformin ID-LC (Intermediate-dose, Long Course) vs SPRY: Metformin HD-SC (High-dose, Short Course) vs SPRY: Metformin HD-IC (High-dose, Intermediate Course) vs SPRY: Placebo; All intervention groups were collapsed into one group and compared with placebo. Patients were compared whether they were discharged home or other; Test type: Superiority; p = 0.72, Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.52 to 1.56]

15. Secondary Outcome: In Hospital Mortality
Time Frame: as for outcome 9
Population: Participants were analyzed using intention-to-trial analysis. Participants that did not undergo an operation were excluded. No in-hospital mortalities were observed and hence no statistical analysis was performed
Measure: Count of Participants; unit: Participants
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
Number analyzed (Participants) | 36 | 20 | 5 | 35 | 19 | 8 | 38 | 23 | 0 | 98
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time the participant is prescribed the study drug until 90 days after surgery.
Description: There is a category with no participants. The total number of participants at risk is different here because adverse events were monitored for all patients while the measure outcomes were only reported for participants that underwent an operation.
  The numbers from this outcome will never match the numbers from outcome 13 since the reporting description is different. e.i a participant can have an AE in multiple systems but are all unrelated; will be counted here several times but there once.
Arm/Group | SPRY: Metformin LD-SC (Low-dose, Short Course) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) | SPRY: Metformin LD-LC (Low-dose, Long Course) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) | SPRY: Metformin HD-SC (High-dose, Short Course) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) | SPRY: Metformin HD-LC (High-dose, Long Course) | SPRY: Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/20 | 0/5 | 1/39 | 0/19 | 0/8 | 0/40 | 0/26 | 0/0 | 0/106
Serious Adverse Events (participants affected / at risk) | 11/39 | 5/20 | 2/5 | 10/39 | 6/19 | 2/8 | 12/40 | 4/26 | 0/0 | 12/106
Other Adverse Events (participants affected / at risk) | 10/39 | 5/20 | 2/5 | 9/39 | 5/19 | 2/8 | 11/40 | 3/26 | 0/0 | 10/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPRY: Metformin LD-SC (Low-dose, Short Course) (N=39) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) (N=20) | SPRY: Metformin LD-LC (Low-dose, Long Course) (N=5) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) (N=39) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) (N=19) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) (N=8) | SPRY: Metformin HD-SC (High-dose, Short Course) (N=40) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) (N=26) | SPRY: Metformin HD-LC (High-dose, Long Course) (N=0) | SPRY: Placebo (N=106)
From time of prescription until 90 days after surgery (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (General disorders) | 4 (5) | 2 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | NA | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | NA | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | NA | 2 (3) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | NA | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Gastrointestinal disorders) | 7 (15) | 4 (4) | 1 (1) | 4 (6) | 5 (9) | 0 (0) | 6 (12) | 3 (3) | NA | 6 (6) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPRY: Metformin LD-SC (Low-dose, Short Course) (N=39) | SPRY: Metformin LD-IC (Low-dose, Intermediate Course) (N=20) | SPRY: Metformin LD-LC (Low-dose, Long Course) (N=5) | SPRY: Metformin ID-SC (Intermediate-dose, Short Course) (N=39) | SPRY: Metformin ID-IC (Intermediate-dose, Intermediate Course) (N=19) | SPRY: Metformin ID-LC (Intermediate-dose, Long Course) (N=8) | SPRY: Metformin HD-SC (High-dose, Short Course) (N=40) | SPRY: Metformin HD-IC (High-dose, Intermediate Course) (N=26) | SPRY: Metformin HD-LC (High-dose, Long Course) (N=0) | SPRY: Placebo (N=106)
Time of prescription of study drug until 90 days after surgery (Gastrointestinal disorders) | 7 (15) | 4 (4) | 1 (1) | 4 (6) | 5 (9) | 0 (0) | 6 (12) | 3 (3) | NA | 6 (6) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription of study drug until 90 days after surgery (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (General disorders) | 4 (5) | 2 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | NA | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0)
Time of prescription until 90 days after surgery (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | NA | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription until 90 days after surgery (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | NA | 2 (3) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription of study drug until 90 days after surgery (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription of study drug until 90 days after surgery (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription of study drug until 90 days after surgery (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | NA | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription of study drug until 90 days after surgery (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription of study drug until 90 days after surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Time of prescription of study drug until 90 days after surgery (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term

LIMITATIONS AND CAVEATS:
Recruitment was terminated early and was limited by the COVID-19 pandemic, as such the study is underpowered and could not meet its set goals. No patients fell in the high dose long course group since no participants were randomized to that group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT03861767/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT03861767/SAP_001.pdf
  • Informed Consent Form (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT03861767/ICF_002.pdf